CLINICAL TRIAL: NCT00919022
Title: Prospective Observational Non-interventional Study of Correlation of Treatment With Androcur, Disease Stage, Testosterone Level, Age With Sexual Function and Erectile Dysfunction (Measured by IIEF-5 Validated Questionnaire)
Brief Title: Androcur Non-interventional Study Among Patients With Carcinoma of the Prostate
Acronym: ANES
Status: Terminated | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer HealthCare AG
Other Study IDs: 14556; AC0910CZ (Other: Company internal)
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: Inoperable Prostate Cancer; Erectile Dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction | interventions — Cyproterone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Cyproterone Acetate (Androcur, BAY94-8367)

INTERVENTIONS:
Drug: Cyproterone Acetate (Androcur, BAY94-8367) — Patients in regular clinical practice receiving Androcur according to local drug information

SUMMARY:
Cyproterone acetate (CPA) is a steroidal antiandrogen which has affinity with progesterone and with glucocorticoid receptors. Cyproterone acetate is long-term proven effective treatment of inoperable carcinoma of the prostate.

Sexual functions remain very important in men with prostate cancer. However sexual functions are deteriorating fast with course of the disease. The influence of CPA on sexual functions remains controversial. IIEF-5 erectile dysfunction questionnaire is currently widely used validated simple scoring system for diagnosing of erectile dysfunction and belongs to most used systems in Czech Republic. At present there are no data on CPA influence on IIEF-5 scored erectile dysfunction within the use of its indication in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males > 18 years previously untreated with Androcur.
* No contraindication to Androcur.

Exclusion Criteria:

* Liver diseases, malignant liver tumours and wasting diseases (except for carcinoma of the prostate). A history of or existing thrombosis or embolism. Severe chronic depression. Hypersensitivity to cyproterone. Cyproterone acetate in previous therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random sample of cancer patients visiting oncologist or urologist ambulance who are suitable for standard Cyproterone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2009-08; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Correlation of treatment with Androcur (concomitant treatment), disease stage, testosterone level, age with erectile dysfunction (measured by IIEF-5 validated questionnaire) | 6 months

SECONDARY OUTCOMES:
Correlation of PSA level and erectile dysfunction | 6 months
Sexual activity of Czech patients with inoperable prostate cancer | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Czechia